CLINICAL TRIAL: NCT03858621
Title: Comparison of Postoperative Nociception Outcomes Between NOL - Guided and Standard Intraoperative Analgesia Based on Fentanyl in Patients Undergoing Elective Surgery With General Anesthesia
Brief Title: Comparison of Postoperative Nociception Between NOL-guided and Standard Intraoperative Analgesia Based on Fentanyl
Acronym: NOLFentanyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Victor Contreras, MSN (Other)
Responsible Party: Sponsor-Investigator, Victor Contreras, MSN, Co-Investigador, Pontificia Universidad Catolica de Chile
Organization: Pontificia Universidad Catolica de Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 180522017; FONDECYT Iniciacion (Other Grant/Funding Number: 11180674)
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative; Opioid Use; Nociceptive Pain; Postoperative Pain; Anesthesia; Allodynia; Analgesics, Opioid
Keywords: pain; Postoperative Pain; fentanyl; Nociceptive monitoring index
MeSH Terms: conditions — Pain, Postoperative; Nociceptive Pain; Hyperalgesia; Pain

STUDY DESIGN:
Intervention Model Description: 2 groups of patients. Randomization into group fentanyl NOL-guided vs fentanyl standard according to randomization list for a total number of 100 patients.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization into group fentanyl NOL-guided vs fentanyl standard will be done prior to the entrance in the OR, the day of the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fentanyl NOL guided (Experimental): A bolus of 2 mcg/kg IV Fentanyl will be given at the induction of the anesthesia. A bolus of 0,5 - 1 mcg/kg IV Fentanyl will be given at the time of incision and during surgery following a predeterminate NOL index + heart rate + mean arterial blood pressure variations.
  Interventions: Drug: fentanyl NOL guided
- fentanyl standard analgesia (No Intervention): A bolus of 2 mcg/kg IV Fentanyl will be given at the induction of the anesthesia. A bolus of 0,5 - 1 mcg/kg IV Fentanyl will be given at the time of incision and during surgery following the heart rate and mean arterial blood pressure variations.

INTERVENTIONS:
Drug: fentanyl NOL guided — Intervention is NOL monitoring in this group that will help to guide intravenous administration of fentanyl during surgery.
  Other Names: NOL analgesia guided fentanyl administration
  Arms: fentanyl NOL guided

SUMMARY:
Pain is defined as an unpleasant sensory and emotional conscious experience, associated with actual or potential tissue damage. Nociception is the sympathetic response to noxious stimuli during unconsciousness. The appearance of different forms of chronic pain results from sensitization of both peripheral and central neural circuits of pain, which involves inflammatory mechanisms both at a systemic level and specifically in the peripheric and central nervous system, as observed through elevation of specific neuroinflammatory mediators, such as MCP-1, IL-1, IL-1b, and IL-10. Clinically, this sensitization expresses as hyperalgesia and allodynia, which increase postoperative pain and morbidity, but also induce permanent modifications in the nociceptive system. These effects may be ameliorated by adequately adjusting intraoperative analgesia through use of nociception/analgesia balance monitors, of which Nociception Level Index (NOL) shows convenient characteristics and promising results from previous studies.

Objectives: The goal of our study is to assess the utility of NOL index monitoring against standard care for Fentanyl-based analgesia by measuring postoperative pain, sensorial thresholds and inflammatory markers related to nociception.

Hypothesis: The use of NOL index to guide the intraoperative analgesia will produce less postoperative pain, hyperalgesia, allodynia, and neuroinflammation.

DETAILED DESCRIPTION:
Methodology: In this RCT double-blinded study will invite to 100 patients aged between 18 and 50 years admitted for elective surgery that is planned to require general anesthesia, with fentanyl as the opioid of choice for intraoperative analgesia.

Each patient will be randomly allocated to one of two groups: the intervention group will be provided intraoperative analgesia guided by NOL values (n=50), and the control group will be provided standard intraoperative analgesia (n=50). To account for inter-personal variability, the NOL threshold value associated with nociceptive stimulation will be assessed on each patient at baseline condition with the Quantitative Sensory Testing (QST) and neuroinflammatory mediators MCP-1, IL-1, IL-1b, and IL-10 will be measured pre- and post-surgery in both groups. Opioid consumption and AVS will be assessed during the stay at the post-surgical care unit as a measurement of post-operative pain and will follow them until three months after surgery.

Statistical Analysis: Results will be expressed as means (±SD) or numbers (%). When indicated, 95% confidence interval (CI) will be calculated. A p-value < 0.05 will be considered statistically significant.

Differences between groups on post-surgical opioid consumption, Δz-score of QST measurements, and serum biomarkers level will be analyzed with Student's T-test for unpaired samples. For analysis purposes, VAS scores will be grouped into three distinct categories: Mild (0-3), Moderate (4-6) and Severe (7-10) pain. Differences between groups will be analyzed with Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Elective abdominal surgery without a neuraxial block.
* Over 2 horas.
* Body Mass Index 18 - 30 kg/m2

Exclusion Criteria:

* Cardiac surgery
* Cardiopathy
* Arrhythmia or use of pacemakers.
* Chronic Kidney disease (Plasma Crea >1 mg/dL).
* Allergic to drugs of this study.
* Opioids or Non-inflammatory drugs over 5 days for two weeks before surgery.
* Neuropathies and dysautonomias.
* Beta-blockers and other drugs that act at the level of the sympathetic system the month prior to surgery.
* Chemotherapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Consumption of IV fentanyl intra-operative in the NOL-guided group compared to the standard group. | Intra-operative
  Total consumption of fentanyl in mcg.
Consumption of opioid in the early postoperative in the NOL-guided group compared to the standard group. | Postoperative Unit (2 hours)
  Total consumption of morphine in mg.

SECONDARY OUTCOMES:
Pain measured by Visual Analog Scale (VAS) in the NOL-guided group compared to the standard group. | Postoperative Unit (Every 30 minutes per 2 hours)
  Visual Analog Scale 0 to 10. 0 = no pain. 10 = worse pain Values to find out is less than 5-6
Sensorial thresholds in the NOL-guided group compared to the standard group. | Postoperative Unit (2 hours)
  QST (Quantitative Sensory Testing) is a valuable method for diagnosing peripheral nervous system disorders.
  1. Thermal Testing
  2. Mechanical test threshold
  3. Mechanical pain threshold
  4. Wind-up phenomenon
  5. Vibration detection threshold
  6. Pressure pain threshold
Pain Management Satisfaction in the NOL-guided group compared to the standard group. | Postoperative Unit (2 hours)
  Pain Management Satisfaction Scale
  1 to 5. 1 = Not satisfied at all. 5 = Completly satisfied One question
Pain Management Satisfaction in the NOL-guided group compared to the standard group. | Postoperative (6 hours)
  Pain Management Satisfaction Scale
  1 to 5. 1 = Not satisfied at all. 5 = Completly satisfied One question
Pain Management Satisfaction in the NOL-guided group compared to the standard group. | Postoperative (12 hours)
  Pain Management Satisfaction Scale
  1 to 5. 1 = Not satisfied at all. 5 = Completly satisfied One question
Inflammatory markers in the NOL-guided group compared to the standard group. | Postoperative (0 hours)
  Concentration in plasma of: MCP1 (pg/mL) , IL6 (pg/mL) , IL1b (pg/mL), IL10 (pg/mL)
Inflammatory markers in the NOL-guided group compared to the standard group. | Postoperative (6 hours)
  Concentration in plasma of: MCP1 (pg/mL) , IL6 (pg/mL) , IL1b (pg/mL), IL10 (pg/mL)
Inflammatory markers in the NOL-guided group compared to the standard group. | Postoperative (12 hours)
  Concentration in plasma of: MCP1 (pg/mL) , IL6 (pg/mL) , IL1b (pg/mL), IL10 (pg/mL)
Persistent pain at three months in the NOL-guided group compared to the standard group. | 3 months after surgery
  Brief Pain Inventory by telephone call

CONTACTS AND LOCATIONS:
Overall Officials: VICTOR CONTRERAS, MSN, Study Director — Research Profesor
Locations (1):
- Victor Contreras, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gandhi K, Heitz JW, Viscusi ER. Challenges in acute pain management. Anesthesiol Clin. 2011 Jun;29(2):291-309. doi: 10.1016/j.anclin.2011.04.009. PMID 21620344
- [Result] Baliki MN, Apkarian AV. Nociception, Pain, Negative Moods, and Behavior Selection. Neuron. 2015 Aug 5;87(3):474-91. doi: 10.1016/j.neuron.2015.06.005. PMID 26247858
- [Result] Katz J, Seltzer Z. Transition from acute to chronic postsurgical pain: risk factors and protective factors. Expert Rev Neurother. 2009 May;9(5):723-44. doi: 10.1586/ern.09.20. PMID 19402781
- [Result] Argoff CE. Recent management advances in acute postoperative pain. Pain Pract. 2014 Jun;14(5):477-87. doi: 10.1111/papr.12108. Epub 2013 Aug 15. PMID 23945010